CLINICAL TRIAL: NCT03660618
Title: LSFG-SKIN, Laser Speckle Flowgraphy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was stopped 3/2/18 as the company who supported the device went out of business and requested the device be returned. Only 1 control subject was tested, no analyzable data.
Sponsor: Randy Kardon (Other)
Responsible Party: Sponsor-Investigator, Randy Kardon, Randy Kardon M.D. Ph.D Professor and Director of Neuro-ophthalmology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201702725
Record Dates: First submitted 2018-07-12; First posted 2018-09-06 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Heart Failure; Vascular Ischemia; Burns; Chemotherapy Effect; Radiation Injuries; Uveitis; Scleritis; Multiple Sclerosis; Autonomic Neuropathy; Stroke; Intracranial Hemorrhages; TIA; Migraine; Headache; Pain
Keywords: perfusion; inflammatory; ischemia; lesions; neuropathy; burns; cancer; stroke
MeSH Terms: conditions — Hypertension; Heart Failure; Burns; Radiation Injuries; Uveitis; Scleritis; Multiple Sclerosis; Stroke; Intracranial Hemorrhages; Migraine Disorders; Headache; Pain; Ischemia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Clinic Subjects (Other): cardiology subjects, dermatology subjects, endocrine subjects, neurology subjects, psychiatry subjects, surgery subjects, ophthalmology subjects.
  Interventions: Device: laser speckle flowgraphy

INTERVENTIONS:
Device: laser speckle flowgraphy — blood flow state of the skin as real time two dimensional image

SUMMARY:
The purpose of this project is to quantify normal and abnormal skin blood flow regionally in different areas of the body(face, extremities, over burns and wounds) at baseline and over time in response to treatment or environmental changes, such as temperature, light and pressure.

DETAILED DESCRIPTION:
Laser speckle skin blood flow (LSFG-SKIN) will be recorded in normal subjects and in patients with disorders affecting skin capillary perfusion, which may include cardiovascular disorders, dermatologic disorders, skin wounds, ocular disorders, psychiatric disorders, and neurologic disorders.

ELIGIBILITY:
Inclusion Criteria:

Controls

●Healthy normal control subjects ages 18-90

Cardiology Subjects

* Ages 18-90
* History of dysrhythmia, heart failure, cardiac ischemia, hypertension, peripheral vascular disease

Dermatology Subjects

* Ages 18-90
* History of inflammatory and cancerous lesions

Endocrine Subjects

* Ages 18-90
* History of diabetes, thyroid disease

Neurology Subjects

* Ages 18-90
* History of dementia, headaches, Parkinson's, light sensitivity, stroke, TIA, multiple sclerosis

Psychiatry Subjects

* Ages 18-90
* History of bipolar, schizophrenia, anxiety, depression

Surgery Subjects

* Ages 18-90
* History of skin wounds(trauma, chemotherapy, radiation), thermal burns, or plastic and reconstructive surgical procedures.

Ophthalmology Subjects

* Ages 18-90
* History of ocular disorders caused by hypo perfusion or inflammatory disorders

Exclusion Criteria:

Controls

* Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.
* Angle closure glaucoma

Cardiology Subjects

* Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.
* Angle closure glaucoma

  3. Dermatology Subjects
* Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.
* Angle closure glaucoma

Endocrine Subjects

* Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.
* Angle closure glaucoma

Neurology Subjects

* Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.
* Angle closure glaucoma

Psychiatry Subjects

* Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.
* Angle closure glaucoma

Surgery Subjects

* Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.
* Angle closure glaucoma

Ophthalmology Subjects

* Cataract or media opacity that would degrade the imaging of the retina. Mild cataracts are okay.
* Angle closure glaucoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Department of Ophthalmology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinic Subjects
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: female
Arm/Group | Clinic Subjects
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Imaging Blood Flow
Description: Imaging blood flow in the tissue is of major importance in the clinical environment
Time Frame: One visit
Population: One subject tested before device had to be returned due to company going out of business. Data was not measurable and no repeat testing was possible as device was returned.
Arm/Group | Clinic Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 5 months.
Description: No adverse events occurred.
Arm/Group | Clinic Subjects
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination due to company going out of business, requested device be returned. No other companies supported this type of device. Early termination lead to only 1 subject enrolled, no analyzable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT03660618/Prot_000.pdf